CLINICAL TRIAL: NCT03580616
Title: Tolerability and Efficacy of L-Serine in Patients With Amyotrophic Lateral Sclerosis: A Phase IIa Study
Brief Title: Tolerability and Efficacy of L-Serine in Patients With Amyotrophic Lateral Sclerosis (ALS)
Acronym: ALS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated by the IRB due to continued noncompliance.
Sponsor: Elijah W. Stommel (Other)
Collaborators: Brain Chemistry Labs (Other)
Responsible Party: Sponsor-Investigator, Elijah W. Stommel, Staff Physician, Neurology, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D18095
Record Dates: First submitted 2018-06-26; First posted 2018-07-09 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Serine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- L-Serine (Experimental): L-Serine 15 grams orally twice a day as tolerated for 6 months
  Interventions: Drug: L-Serine

INTERVENTIONS:
Drug: L-Serine — L-Serine is a naturally occurring dietary amino acid. It is abundant in soy products, some edible seaweeds, sweet potatoes, eggs and meat.

SUMMARY:
The purpose of this study is to determine the tolerability of L-Serine oral doses for ALS patients and assess preliminary indications of efficacy

DETAILED DESCRIPTION:
All patients will receive the same dose of the study treatment over 6 months. For each participant the study will last approximately one year with follow up visits after the treatment period of 6 months is completed. The visits will include blood draws, vital sign checks, neurological and physical exams, pulmonary testing with forced vital capacity (FVC), and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable or definite ALS
* ALSFRS-R score >25 and FVC score ≥ 60% predicted
* If currently taking Riluzole and/or Edaravone/Radicava must be on stable dose for 3 months prior to Baseline/Screening. If the dosing has not been stable for 3 months prior to Baseline/Screening or if stopped due to an adverse event, the waiting period off the medication will be 7 days. If not on either of these medications may start if desired either or both medications after enrollment into study.

Exclusion Criteria:

* Diagnosis of probable or definite ALS more than 3 years prior to study enrollment
* Diagnosis or previous history of ischemic stroke, brain tumor, uncontrolled diabetes, renal insufficiency, or severe hypertension.
* Diagnosis or previous history of comorbid progressive neurodegenerative disease such as Alzheimer's disease, Parkinson's disease, Lewy Body disease, Pick's disease, Huntington's disease, Progressive Supranuclear palsy. ALS patients diagnosed with frontotemporal dementia will not be excluded from this study.
* Diagnosis or previous history of symptomatic peripheral neuropathy. Patients with findings of peripheral neuropathy on electrodiagnostic tests only but no clinical symptoms at the time of enrollment are eligible.
* Undergoing any chemotherapy or radiation therapy for any cancer
* Any medical condition likely to interfere with the conduct of the trial or survival of the patient during this study period
* Pregnant women or women who are breast feeding
* Has taken L-Serine supplement within 30 days prior to start of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elijah W Stommel, MD,PHD, Principal Investigator — Dartmouth-Htichcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Background] Abe K, Itoyama Y, Sobue G, Tsuji S, Aoki M, Doyu M, Hamada C, Kondo K, Yoneoka T, Akimoto M, Yoshino H; Edaravone ALS Study Group. Confirmatory double-blind, parallel-group, placebo-controlled study of efficacy and safety of edaravone (MCI-186) in amyotrophic lateral sclerosis patients. Amyotroph Lateral Scler Frontotemporal Degener. 2014 Dec;15(7-8):610-7. doi: 10.3109/21678421.2014.959024. Epub 2014 Oct 6. PMID 25286015
- [Background] Andrew AS, Caller TA, Tandan R, Duell EJ, Henegan PL, Field NC, Bradley WG, Stommel EW. Environmental and Occupational Exposures and Amyotrophic Lateral Sclerosis in New England. Neurodegener Dis. 2017;17(2-3):110-116. doi: 10.1159/000453359. Epub 2017 Jan 26. PMID 28122372
- [Background] Brannath W, Burger HU, Glimm E, Stallard N, Vandemeulebroecke M, Wassmer G. Comments on the draft guidance on "adaptive design clinical trials for drugs and biologics" of the U.S. Food and Drug Administration. J Biopharm Stat. 2010 Nov;20(6):1125-31. doi: 10.1080/10543406.2010.514453. PMID 21058108
- [Background] Banack SA, Murch SJ, Cox PA. Neurotoxic flying foxes as dietary items for the Chamorro people, Marianas Islands. J Ethnopharmacol. 2006 Jun 15;106(1):97-104. doi: 10.1016/j.jep.2005.12.032. Epub 2006 Feb 7. PMID 16457975
- [Background] Braak H, Braak E. Staging of Alzheimer's disease-related neurofibrillary changes. Neurobiol Aging. 1995 May-Jun;16(3):271-8; discussion 278-84. doi: 10.1016/0197-4580(95)00021-6. PMID 7566337
- [Background] Caller TA, Andrews A, Field NC, Henegan PL, Stommel EW. The Epidemiology of Amyotrophic Lateral Sclerosis in New Hampshire, USA, 2004-2007. Neurodegener Dis. 2015;15(4):202-6. doi: 10.1159/000374117. Epub 2015 Apr 16. PMID 25896575
- [Background] Canu N, Ciotti MT, Pollegioni L. Serine racemase: a key player in apoptosis and necrosis. Front Synaptic Neurosci. 2014 Apr 21;6:9. doi: 10.3389/fnsyn.2014.00009. eCollection 2014. PMID 24795622
- [Background] Cox PA, Banack SA, Murch SJ. Biomagnification of cyanobacterial neurotoxins and neurodegenerative disease among the Chamorro people of Guam. Proc Natl Acad Sci U S A. 2003 Nov 11;100(23):13380-3. doi: 10.1073/pnas.2235808100. PMID 14612559
- [Background] Cox PA, Davis DA, Mash DC, Metcalf JS, Banack SA. Dietary exposure to an environmental toxin triggers neurofibrillary tangles and amyloid deposits in the brain. Proc Biol Sci. 2016 Jan 27;283(1823):20152397. doi: 10.1098/rspb.2015.2397. PMID 26791617
- [Background] de Koning TJ. Treatment with amino acids in serine deficiency disorders. J Inherit Metab Dis. 2006 Apr-Jun;29(2-3):347-51. doi: 10.1007/s10545-006-0269-0. PMID 16763900
- [Background] Desai JR, Bowen EA, Danielson MM, Allam RR, Cantor MN. Creation and implementation of a historical controls database from randomized clinical trials. J Am Med Inform Assoc. 2013 Jun;20(e1):e162-8. doi: 10.1136/amiajnl-2012-001257. Epub 2013 Feb 28. PMID 23449762
- [Background] Dunlop RA, Cox PA, Banack SA, Rodgers KJ. The non-protein amino acid BMAA is misincorporated into human proteins in place of L-serine causing protein misfolding and aggregation. PLoS One. 2013 Sep 25;8(9):e75376. doi: 10.1371/journal.pone.0075376. eCollection 2013. PMID 24086518
- [Background] Dunlop RA, Powell J, Guillemin GJ, Cox PA. Mechanisms of L-Serine Neuroprotection in vitro Include ER Proteostasis Regulation. Neurotox Res. 2018 Jan;33(1):123-132. doi: 10.1007/s12640-017-9829-3. Epub 2017 Nov 2. PMID 29098664
- [Background] Dunlop RA, Powell JT, Metcalf JS, Guillemin GJ, Cox PA. L-Serine-Mediated Neuroprotection Includes the Upregulation of the ER Stress Chaperone Protein Disulfide Isomerase (PDI). Neurotox Res. 2018 Jan;33(1):113-122. doi: 10.1007/s12640-017-9817-7. Epub 2017 Oct 3. PMID 28975502
- [Background] Fiandaca MS, Kapogiannis D, Mapstone M, Boxer A, Eitan E, Schwartz JB, Abner EL, Petersen RC, Federoff HJ, Miller BL, Goetzl EJ. Identification of preclinical Alzheimer's disease by a profile of pathogenic proteins in neurally derived blood exosomes: A case-control study. Alzheimers Dement. 2015 Jun;11(6):600-7.e1. doi: 10.1016/j.jalz.2014.06.008. Epub 2014 Aug 15. PMID 25130657
- [Background] Garofalo K, Penno A, Schmidt BP, Lee HJ, Frosch MP, von Eckardstein A, Brown RH, Hornemann T, Eichler FS. Oral L-serine supplementation reduces production of neurotoxic deoxysphingolipids in mice and humans with hereditary sensory autonomic neuropathy type 1. J Clin Invest. 2011 Dec;121(12):4735-45. doi: 10.1172/JCI57549. PMID 22045570
- [Background] Goetzl EJ, Boxer A, Schwartz JB, Abner EL, Petersen RC, Miller BL, Kapogiannis D. Altered lysosomal proteins in neural-derived plasma exosomes in preclinical Alzheimer disease. Neurology. 2015 Jul 7;85(1):40-7. doi: 10.1212/WNL.0000000000001702. Epub 2015 Jun 10. PMID 26062630
- [Background] Hirtz D, Thurman DJ, Gwinn-Hardy K, Mohamed M, Chaudhuri AR, Zalutsky R. How common are the "common" neurologic disorders? Neurology. 2007 Jan 30;68(5):326-37. doi: 10.1212/01.wnl.0000252807.38124.a3. PMID 17261678
- [Background] Kabashi E, Valdmanis PN, Dion P, Spiegelman D, McConkey BJ, Vande Velde C, Bouchard JP, Lacomblez L, Pochigaeva K, Salachas F, Pradat PF, Camu W, Meininger V, Dupre N, Rouleau GA. TARDBP mutations in individuals with sporadic and familial amyotrophic lateral sclerosis. Nat Genet. 2008 May;40(5):572-4. doi: 10.1038/ng.132. Epub 2008 Mar 30. PMID 18372902
- [Background] Kaufmann P, Levy G, Thompson JL, Delbene ML, Battista V, Gordon PH, Rowland LP, Levin B, Mitsumoto H. The ALSFRSr predicts survival time in an ALS clinic population. Neurology. 2005 Jan 11;64(1):38-43. doi: 10.1212/01.WNL.0000148648.38313.64. PMID 15642901
- [Background] Logroscino G, Traynor BJ, Hardiman O, Chio A, Mitchell D, Swingler RJ, Millul A, Benn E, Beghi E; EURALS. Incidence of amyotrophic lateral sclerosis in Europe. J Neurol Neurosurg Psychiatry. 2010 Apr;81(4):385-90. doi: 10.1136/jnnp.2009.183525. Epub 2009 Aug 25. PMID 19710046
- [Background] Mehta P, Kaye W, Bryan L, Larson T, Copeland T, Wu J, Muravov O, Horton K. Prevalence of Amyotrophic Lateral Sclerosis - United States, 2012-2013. MMWR Surveill Summ. 2016 Aug 5;65(8):1-12. doi: 10.15585/mmwr.ss6508a1. PMID 27490513
- [Background] Metcalf JS, Dunlop RA, Powell JT, Banack SA, Cox PA. L-Serine: a Naturally-Occurring Amino Acid with Therapeutic Potential. Neurotox Res. 2018 Jan;33(1):213-221. doi: 10.1007/s12640-017-9814-x. Epub 2017 Sep 19. PMID 28929385
- [Background] Metcalf JS, Lobner D, Banack SA, Cox GA, Nunn PB, Wyatt PB, Cox PA. Analysis of BMAA enantiomers in cycads, cyanobacteria, and mammals: in vivo formation and toxicity of D-BMAA. Amino Acids. 2017 Aug;49(8):1427-1439. doi: 10.1007/s00726-017-2445-y. Epub 2017 Jun 15. PMID 28620737
- [Background] Murch SJ, Cox PA, Banack SA. A mechanism for slow release of biomagnified cyanobacterial neurotoxins and neurodegenerative disease in Guam. Proc Natl Acad Sci U S A. 2004 Aug 17;101(33):12228-31. doi: 10.1073/pnas.0404926101. Epub 2004 Aug 4. PMID 15295100
- [Background] Phukan J, Elamin M, Bede P, Jordan N, Gallagher L, Byrne S, Lynch C, Pender N, Hardiman O. The syndrome of cognitive impairment in amyotrophic lateral sclerosis: a population-based study. J Neurol Neurosurg Psychiatry. 2012 Jan;83(1):102-8. doi: 10.1136/jnnp-2011-300188. Epub 2011 Aug 11. PMID 21836033
- [Background] Polman CH, Reingold SC, Barkhof F, Calabresi PA, Clanet M, Cohen JA, Cutter GR, Freedman MS, Kappos L, Lublin FD, McFarland HF, Metz LM, Miller AE, Montalban X, O'Connor PW, Panitch H, Richert JR, Petkau J, Schwid SR, Sormani MP, Thompson AJ, Weinshenker BG, Wolinsky JS. Ethics of placebo-controlled clinical trials in multiple sclerosis: a reassessment. Neurology. 2008 Mar 25;70(13 Pt 2):1134-40. doi: 10.1212/01.wnl.0000306410.84794.4d. PMID 18362273
- [Background] Ringholz GM, Appel SH, Bradshaw M, Cooke NA, Mosnik DM, Schulz PE. Prevalence and patterns of cognitive impairment in sporadic ALS. Neurology. 2005 Aug 23;65(4):586-90. doi: 10.1212/01.wnl.0000172911.39167.b6. PMID 16116120
- [Background] Splawinski J, Kuzniar J. Clinical trials: active control vs placebo--what is ethical? Sci Eng Ethics. 2004 Jan;10(1):73-9. doi: 10.1007/s11948-004-0065-x. PMID 14986774
- [Background] Thall PF, Simon RM, Estey EH. Bayesian sequential monitoring designs for single-arm clinical trials with multiple outcomes. Stat Med. 1995 Feb 28;14(4):357-79. doi: 10.1002/sim.4780140404. PMID 7746977
- [Background] Thompson AG, Gray E, Heman-Ackah SM, Mager I, Talbot K, Andaloussi SE, Wood MJ, Turner MR. Extracellular vesicles in neurodegenerative disease - pathogenesis to biomarkers. Nat Rev Neurol. 2016 Jun;12(6):346-57. doi: 10.1038/nrneurol.2016.68. Epub 2016 May 13. PMID 27174238
- [Background] Viele K, Berry S, Neuenschwander B, Amzal B, Chen F, Enas N, Hobbs B, Ibrahim JG, Kinnersley N, Lindborg S, Micallef S, Roychoudhury S, Thompson L. Use of historical control data for assessing treatment effects in clinical trials. Pharm Stat. 2014 Jan-Feb;13(1):41-54. doi: 10.1002/pst.1589. Epub 2013 Aug 5. PMID 23913901
- [Background] Wheaton MW, Salamone AR, Mosnik DM, McDonald RO, Appel SH, Schmolck HI, Ringholz GM, Schulz PE. Cognitive impairment in familial ALS. Neurology. 2007 Oct 2;69(14):1411-7. doi: 10.1212/01.wnl.0000277422.11236.2c. PMID 17909153
- [Background] Winston CN, Goetzl EJ, Akers JC, Carter BS, Rockenstein EM, Galasko D, Masliah E, Rissman RA. Prediction of conversion from mild cognitive impairment to dementia with neuronally derived blood exosome protein profile. Alzheimers Dement (Amst). 2016 May 7;3:63-72. doi: 10.1016/j.dadm.2016.04.001. eCollection 2016. PMID 27408937
- [Background] Brooks BR, Miller RG, Swash M, Munsat TL; World Federation of Neurology Research Group on Motor Neuron Diseases. El Escorial revisited: revised criteria for the diagnosis of amyotrophic lateral sclerosis. Amyotroph Lateral Scler Other Motor Neuron Disord. 2000 Dec;1(5):293-9. doi: 10.1080/146608200300079536. No abstract available. PMID 11464847
- [Background] Cedarbaum JM, Stambler N, Malta E, Fuller C, Hilt D, Thurmond B, Nakanishi A. The ALSFRS-R: a revised ALS functional rating scale that incorporates assessments of respiratory function. BDNF ALS Study Group (Phase III). J Neurol Sci. 1999 Oct 31;169(1-2):13-21. doi: 10.1016/s0022-510x(99)00210-5. PMID 10540002
- [Background] Levine TD, Miller RG, Bradley WG, Moore DH, Saperstein DS, Flynn LE, Katz JS, Forshew DA, Metcalf JS, Banack SA, Cox PA. Phase I clinical trial of safety of L-serine for ALS patients. Amyotroph Lateral Scler Frontotemporal Degener. 2017 Feb;18(1-2):107-111. doi: 10.1080/21678421.2016.1221971. Epub 2016 Sep 2. PMID 27589995

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Routine monitoring revealed major noncompliance that was not adequately addressed by the Sponsor-Investigator. Subsequently, the study was terminated by the Institutional Review Board (IRB). The IRB determined these deviations compromised the integrity of the data. Furthermore, the study data collected have been deemed unreliable due to issues related to the study's conduct.
Groups:
- L-Serine: Participants who provided consent.
Period: Overall Study
Arm/Group | L-Serine
Started (Provided Consent) | 43
Was Determined Eligible at Screening Visit | 37
Included in Interim Analysis | 28
Completed | 0 (Completed all visits and phone calls as described by the protocol.)
Not Completed | 43

BASELINE CHARACTERISTICS:
Population: Participants determined to be eligible at screening visit
Groups:
- L-Serine: Participants determined to be eligible at screening visit
Arm/Group | L-Serine
Number analyzed (Participants) | 37
Age, Customized [Count of Participants; unit: Participants]
  50 - 59 years | 14
  60 - 69 years | 12
  70 - 79 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 35
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Dose Tolerability Based on Subject Reporting
Description: Tolerability was based off of participant self-reported GI symptoms at any time during their participation.
Time Frame: From baseline through when participants withdrew from study or up to 48 weeks
Population: Routine monitoring revealed major noncompliance that was not adequately addressed by the Sponsor-Investigator. Subsequently, the study was terminated by the Institutional Review Board (IRB). The IRB determined these deviations compromised the integrity of the data. Furthermore, the study data collected have been deemed unreliable due to issues related to the study's conduct.
Measure: Count of Participants; unit: Participants
Arm/Group | L-Serine
Number analyzed (Participants) | 37
Participants
  Diarrhea | 7
  Bowel Obstruction | 1
  Nausea | 8

2. Secondary Outcome: Mean ALS Functional Rating Scale - Revised (ALSFRS-R) Score
Description: Amyotrophic lateral sclerosis functional rating scale-revised version (ALSFRS-R) is used to determine patients' assessments of their capability and independence in 12 functional activities. All 12 activities are relevant in ALS and each is scored between 0 (no function at all) and 4 (normal function). Thus the overall score for this measure can range from 0 to 48, with higher scores indicating more normal function.
Time Frame: Baseline through 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Mean score
Groups:
- L-Serine: Participants involved in interim analysis
Arm/Group | L-Serine
Number analyzed (Participants) | 28
Mean score | 28.8732 (5.3734)

3. Secondary Outcome: Efficacy Based on Pulmonary Forced Vital Capacity (FVC) as Measured by Mean Slope Through Time
Time Frame: No data available
Population: Routine monitoring revealed major noncompliance that was not adequately addressed by the Sponsor-Investigator. Subsequently, study was terminated by the Institutional Review Board. The protocol specified that this outcome measure would obtain the slope through time as a measure of efficacy based on FVC. Although raw data for the FVC was collected, these data were not analyzed and slope values were not obtained before study closure. The slope values will never be obtained due to study termination
Arm/Group | L-Serine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The adverse event data was collected from baseline through when participants withdrew from study or up to 48 weeks.
Description: Routine monitoring revealed major noncompliance that was not adequately addressed by the Sponsor-Investigator. Subsequently, the study was terminated by the Institutional Review Board (IRB). The IRB determined these deviations compromised the integrity of the data. Furthermore, the study data collected have been deemed unreliable due to issues related to the study's conduct.
Arm/Group | L-Serine
All-Cause Mortality (participants affected / at risk) | 1/37
Serious Adverse Events (participants affected / at risk) | 12/37
Other Adverse Events (participants affected / at risk) | 31/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-Serine (N=37)
Respiratory Arrest (Cardiac disorders) | 1 (1)
Bowel Obstruction (Gastrointestinal disorders) | 1 (1)
Viral infection and mild rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 1 (1)
Breathing difficulty/Ventilation Issues (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Gastric tube Placement (Surgical and medical procedures) | 2 (2)
Pre-Planned Surgical Procedure (Surgical and medical procedures) | 1 (1)
Worsening weakness and Falls (Musculoskeletal and connective tissue disorders) | 1 (1)
Bimalleolar Fracture with Lateral Subluxation (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-Serine (N=37)
Falls (Musculoskeletal and connective tissue disorders) | 16 (24)
Diarrhea (Gastrointestinal disorders) | 7 (12)
Nausea (Gastrointestinal disorders) | 8 (15)

LIMITATIONS AND CAVEATS:
Routine monitoring revealed major noncompliance that was not adequately addressed by the Sponsor-Investigator. Subsequently, the study was terminated by the Institutional Review Board (IRB). The IRB determined these deviations compromised the integrity of the data. Furthermore, the study data collected have been deemed unreliable due to issues related to the study's conduct.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/16/NCT03580616/Prot_SAP_000.pdf